CLINICAL TRIAL: NCT04604873
Title: The Integrated Support and Palliative in Cancer Day-care Hospital for Patients With Advanced Cancers: Impact on Quality of Life, Care Pathways and Support for Caregivers
Brief Title: The Integrated Support and Palliative in Cancer Day-care Hospital for Patients With Advanced Cancers: Impact on Quality of Life, Care Pathways and Support for Caregivers (HDJ-SPI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IC 2019-08
Record Dates: First submitted 2020-10-20; First posted 2020-10-27 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Cancer, Advanced
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No hospital one day care (No Intervention): No hospital one day care
- Hospital one day care (Other): Hospital one day care
  Interventions: Other: Hospital day care follow-up

INTERVENTIONS:
Other: Hospital day care follow-up — Regular follow up every month in hospital day care
  Arms: Hospital one day care

SUMMARY:
The main objective is to show the impact on the quality of life (QoL) for adults patients with advanced cancer managed in day hospital of integrated palliative care of cancer center (HDJ-SPI).

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥ 18 years old with advanced solid tumor
2. Addressed for the first time to the palliative care team according to current criteria (medico-psycho-social symptoms, progressive risks)
3. With or without anti-cancer treatment
4. With estimated life expectancy of more than 2 months and less than 12 months
5. Able to communicate in French and answer questionnaires
6. Affiliated with a social security system
7. Having signed informed consent, co-signed by the partner if designated by the patient

Exclusion Criteria:

1. Patient with primitive brain tumor or malignant hemopathy
2. Severe psychopathological disorders
3. Pregnant patient or childbearing potential without effective method of birth control
4. Unable to be followed at the cancer center until death
5. Patient deprived of liberty or under guardianship -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Analyse impact of hospital day care in integrated palliative care department on quality of life of adult patients with advanced stage cancer | 12 months
  Analyse impact of hospital day care in integrated palliative care department on quality of life of adult patients with advanced stage cancer
  Outcome shall be evaluated by assessing Survival without quality of life deterioration,measured by EORTC QLQ-C30 scale with monthly evaluation targeting three dimensions :
  global quality of life/ fatigue/ patient emotional state

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Institut Bergonie, Bordeaux
  - Centre Antoine Lacassagne, Nice
  - Institutcurie Paris, Paris
  - INSTITUT CURIE Saint-Cloud, Saint-Cloud
  - Institut de Cancerologie de L'Ouest, Saint-Herblain
  - Centre Paul Strauss, Strasbourg

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific reserach, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).

REFERENCES:
- [Derived] Marret L, Anota A, Waechter L, Laouisset C, Marchal T, Burnod A, Angellier E, Djoumakh OEK, Thebaut C, Bredart A, Dolbeault S, Mino JC, Bouleuc C. Palliative care in day-hospital for advanced cancer patients: a study protocol for a multicentre randomized controlled trial. BMC Palliat Care. 2021 Apr 17;20(1):61. doi: 10.1186/s12904-021-00754-x. PMID 33865379